CLINICAL TRIAL: NCT00003685
Title: A Phase III Trial of Single Versus Fractionated Thoracic Radiation for Palliation of Symptoms in Patients With Non-Small Cell Lung Cancer
Brief Title: Radiation Therapy to Relieve Symptoms in Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC15; CAN-NCIC-SC15 (Other: PDQ); CDR0000066787 (Other: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-05-20 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Fatigue; Lung Cancer; Nausea and Vomiting; Pain; Pulmonary Complications; Quality of Life
Keywords: stage III non-small cell lung cancer; recurrent non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; fatigue; nausea and vomiting; pain; pulmonary complications; quality of life
MeSH Terms: conditions — Fatigue; Lung Neoplasms; Nausea; Vomiting; Pain; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Therapeutics; Analgesia; Radiotherapy

INTERVENTIONS:
Procedure: fatigue assessment and management
Procedure: nausea and vomiting therapy
Procedure: pain therapy
Procedure: quality-of-life assessment
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy may relieve symptoms in patients with non-small cell lung cancer. It is not yet known which regimen of radiation therapy is most effective in relieving symptoms in patients with non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of different regimens of radiation therapy to relieve symptoms in patients who have non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of two schedules of radiotherapy in the palliation of symptoms in patients with non-small cell lung cancer. II. Compare the toxicity of these two regimens in these patients. III. Compare the quality of life and survival of patients treated with these two regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, weight loss in the previous 6 months (no greater than 10% vs greater than 10%), and performance status (ECOG 0 or 1 vs 2 or 3). Patients are randomized to undergo radiotherapy as 5 fractions over 5 days or 1 fraction on 1 day. Quality of life is assessed before treatment, weekly for 5 weeks, and monthly thereafter. Patients are followed weekly for 5 weeks, then every 2 months for 1 year.

PROJECTED ACCRUAL: A total of 210 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven non-small cell lung cancer Squamous cell lung cancer Large cell lung cancer Adenocarcinoma lung cancer Mixture of above Locally advanced disease for which the patient declined aggressive treatment or that is unsuitable for aggressive curative treatment due to at least one of the following: Performance status of ECOG 2 or 3 Otherwise unexplained weight loss greater than 10% in the last 6 months Bulky disease that cannot be irradiated safely to high doses Inability to tolerate chemotherapy Cytologically positive pleural effusion OR Clinically or radiologically proven metastatic disease for which palliative chemotherapy is not planned in the first 38 days after radiotherapy No more than one brain metastasis allowed One of the following symptoms identified as the index symptom: Loss of appetite Nausea Vomiting Cough Coughing up blood Chest pain Shortness of breath Difficulty swallowing Fatigue Must have symptoms related to intrathoracic lung cancer that are amenable to radiation palliation

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: ECOG 0-3 Life expectancy: Greater than 3 months Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Fluent in English or French No loss of sight or other inability to complete questionnaires or diary Not pregnant No concurrent terminal illness No other active malignancy that is causing symptoms or is expected to progress in the next 3 months

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 30 days since prior chemotherapy and failed No planned chemotherapy within 38 days after study treatment Endocrine therapy: Not specified Radiotherapy: No planned laser therapy within 38 days after study treatment Surgery: At least 30 days since prior surgery and failed Other: No planned photodynamic therapy or sclerotherapy within 38 days after study treatment

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 1997-08-01 (Actual); Primary Completion 2001-03 (Actual); Study Completion 2009-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bezjak, MD, MSC, FRCPC, Study Chair — Princess Margaret Hospital, Canada
Locations (21):
- Canada (21):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BC Cancer Agency, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Ottawa Regional Cancer Center - General Division, Ottawa, Ontario
  - Ottawa Regional Cancer Centre - Civic Campus, Ottawa, Ontario
  - Peterborough Oncology Clinic, Peterborough, Ontario
  - Hotel Dieu Hospital - St. Catharines, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bezjak A, Dixon P, Brundage M, Tu D, Palmer MJ, Blood P, Grafton C, Lochrin C, Leong C, Mulroy L, Smith C, Wright J, Pater JL; Clinical Trials Group of the National Cancer Institute of Canada. Randomized phase III trial of single versus fractionated thoracic radiation in the palliation of patients with lung cancer (NCIC CTG SC.15). Int J Radiat Oncol Biol Phys. 2002 Nov 1;54(3):719-28. doi: 10.1016/s0360-3016(02)02989-9. PMID 12377323